CLINICAL TRIAL: NCT06348082
Title: Implementing Mindfulness Practice to Advance Sleep Health Equity Among Black Women
Brief Title: Project Women's Insomnia Sleep Health Equity Study (WISHES)
Acronym: Project WISHES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2000036068; 1R18HS029812-01 (AHRQ)
Record Dates: First submitted 2024-02-07; First posted 2024-04-04 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Insomnia; Sleep Health; Cardiometabolic Health
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Hybrid Type 1 effectiveness/implementation study using a pragmatic randomized controlled trial (RCT) with MBTI and a waitlist control. Participants will be randomly assigned by a computer-generated sequence to either the MBTI or waitlist control in a 1:1 ratio using permuted blocks stratified by age (2 strata: ≤50 or postmenopausal age >51) with random block sizes of 2 or 4 to reduce predictability.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBTI (Experimental): Participants randomized to MBTI group.
  Interventions: Behavioral: Mindfulness-based therapy for insomnia (MBTI)
- Control (No Intervention): Participants randomized to waitlist control group.

INTERVENTIONS:
Behavioral: Mindfulness-based therapy for insomnia (MBTI) — MBTI will be administered in 6 weekly sessions. Session 1 consists of introductions and an overview. Subsequent sessions consist of mindfulness concepts/practice and behavioral strategies for sleep. Each session will begin with guided formal meditation followed by discussion. Mindfulness practice (at home) expectations are 30-45 minutes of meditation/day at least 5 days during the period of the intervention, followed by 20 minutes/day until the final follow-up assessment (at 12 weeks). Mindfulness concepts: Overview of Mindfulness, Mindfulness of the Body, Obstacles to Mindfulness, Working with Difficult Emotions, Cultivating Positive Emotions, Working with Difficult Thoughts, Mindful Interactions.
  Arms: MBTI

SUMMARY:
The purpose of this study is to achieve health and healthcare equity by implementing an equity-focused, mindfulness-based sleep intervention to reduce stress and sleep deficiency-related cardiometabolic disease burden in Black women.

DETAILED DESCRIPTION:
In phases 1 and 2, the investigator will identify multi-level barriers and facilitators to implementing the online mindfulness-based therapy for insomnia (MBTI) through an equity lens using community-engaged research with key stakeholders. The investigators will then develop and refine equity-focused implementation strategies with the community advisory board, comprised of community-based organization members, African Methodist Episcopal Zion Church networks, clinicians, and community health workers (CHWs). In phase 3, the investigators will use a Hybrid Type 1 effectiveness/implementation design with a pragmatic randomized controlled trial with MBTI and a waitlist control in Black women with insomnia. Specialists will assess and address social needs of Black women, and registered nurses will deliver the online MBTI intervention in the community settings. The focus of this registration is phase 3.

The study will contribute to equity-focused implementation science and policy decisions by providing multi-level implementation determinants, equity-relevant metrics, and contextual factors through community-engaged research and evaluation of the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* self-identified Black women
* English speaking
* meet ICSD3 diagnostic criteria for insomnia disorders, defined as difficulty initiating or maintaining sleep that occurs despite adequate opportunity to sleep with at least one associated daytime impairment symptom (ISI > 7)
* additional quantitative insomnia criteria based on research recommendations and the new ICSD3: (a) severity of sleep onset latency or wake time after sleep onset of ≥31 min, (b) occurring ≥3 nights a week, and (c) for ≥ 3 months.

Exclusion Criteria:

* Psychosis or unstable/significant depression, anxiety, or substance abuse under active care (more than 1 monthly mental healthcare visit or requiring more than 1 psychotropic medicine daily)
* significant current practice of any form of meditation (>15min per day)
* obstructive sleep apnea (OSA), restless legs syndrome (RLS), or circadian rhythm related condition (shift worker, use of medication that influence circadian rhythm, e.g., Parkinson's disease)
* active or terminal cancer.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 340 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity | baseline, week 6 and week 12
  Change in Insomnia severity or remission will be assessed using the Insomnia Severity Index (ISI). The ISI is a 7 item survey used to determine insomnia severity. Total score range from 0-28 with cutoffs as follows: no insomnia (0-7), sub-threshold insomnia (8-14), moderate insomnia (15-21), and severe insomnia (22-28). Response to the MBTI on the ISI will be defined as a meaningful change of 7 or more points from baseline, or remission as reduction to a score less than 8.
Change in Perceived Stress | baseline, week 6 and week 12
  Change will be assessed using the Perceived Stress Scale (PSS -10) Total score range from 0-40 with cutoffs as follows: low perceived stress (0-13); moderate perceived stress (14-26); high perceived stress (27-40). Response to the MBTI on the PSS will be defined as a meaningful change of 5 or more points from baseline, or remission as reduction to a score less than 13.
Acceptability of Intervention (AIM) | week 6 and week 12
  Acceptability of the implementation strategy will be assessed using the Acceptability of Intervention measure (AIM). It has 4-items scored on a 5-point Likert scale summed to achieve a total score. Total score range of 0-20. Higher scores indicate more acceptability.
Feasibility of Intervention (FIM) | week 6 and week 12
  Feasibility of the implementation strategy will be assessed using the Acceptability of Intervention measure (FIM). It has 4-items scored on a 5-point Likert scale summed to achieve a total score. Total score range of 0-20. Higher scores indicate higher likelihood of feasibility.
Treatment Fidelity | Weeks 1-6 intervention training sessions
  Fidelity to the MBTI intervention will be scored using The Mindfulness-Based Relapse Prevention Adherence and Competence Scale (MBRP-AC), a treatment fidelity checklist tool for mindfulness interventions. Specifically, staff trained to observe key components of intervention delivery will complete a checklist of items that correspond to each session (n=8) to evaluate the fidelity to the intervention protocol. Summary scores will reflect the higher the percentage of key components checked off, the higher the fidelity to the treatment intervention protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Soohyun Nam, PhD, APRN, ANP-BC, FAHA, FAAN, Principal Investigator — Yale University School of Nursing
Locations (1):
- Yale School of Nursing Biobehavioral Lab, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will publish a number of manuscripts related to the methods, implementation process, and the trial analyses planned for the project. These will be published in a timely fashion as soon as data can be shared. Investigators plan to widely disseminate the findings of this project to the scientific community by presenting the findings at numerous scientific meetings and will make these slide presentations available to the research community. Investigators will also disseminate our scientific products in lay formats (e.g., research briefs, infographics) through our Expert Advisory Board and community partners. Investigators plan to make available the cleaned and completely de-identified datasets and PDF versions of our research forms and research protocol.
Supporting Information: Study Protocol
Time Frame: Data will be available as soon as the trial ends and until 6 years after the completion of the trial
Access Criteria: A data sharing agreement will be required for release of any data. Individuals requesting a copy of study data will need to submit a detailed research plan that includes the purpose of the proposed research, the variables required, the duration of the analysis phase, IRB approval, investigator training in human subjects and other approvals specific to the individual datasets. They will also be required to submit a Data Protection Plan or Institutional Privacy Policy, describing the computing environment in which data will be managed and analyzed and how physical access to computing equipment will be controlled. Data will only be released once all IRB approvals and Human Subjects concerns have been addressed. Data collection instruments, codebooks, and other data documentation will be made available in conjunction with this dataset in a standard format that is readable across a variety of applications and operating system platforms.

REFERENCES:
- [Derived] Nam S, Tong G, Iennaco J, Humphries D, Ordway M, Lee M, Thompson S, Seguinot M, Morales F, Harriot K, Paris N, Bryant KA, Weidner K, Edwards T, Whittemore R. Protocol for a hybrid type 1 effectiveness-implementation study of mindfulness-based therapy for insomnia in Black women. Contemp Clin Trials. 2026 Jan;160:108166. doi: 10.1016/j.cct.2025.108166. Epub 2025 Nov 25. PMID 41308952